CLINICAL TRIAL: NCT02256540
Title: The Effects of Resveratrol and Acute Exercise on Endothelial Function in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 14-0532; UL1TR001082 (NIH); R56HL114073 (NIH)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Estradiol; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo patch - placebo tablets (Placebo Comparator): Postmenopausal women will be given a placebo patch to wear two days prior to exercise visit and a placebo tablet to take the morning of the exercise visit.
  Interventions: Drug: Placebo patch; Dietary Supplement: Placebo
- Placebo patch - Resveratrol tablets (Experimental): Postmenopausal women will be given a placebo patch to wear for two days prior to the exercise visit and a resveratrol tablet (dosed at 250mg) to take the morning of the exercise visit.
  Interventions: Drug: Placebo patch; Dietary Supplement: Resveratrol
- Climara patch - placebo tablets (Active Comparator): Postmenopausal women will be given a transdermal estrogen patch to wear (0.05mg/day) for two days prior to the exercise visit and a placebo tablet to take the morning of the exercise visit.
  Interventions: Drug: Climara; Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Climara
  Other Names: Estradiol transdermal patch
  Arms: Climara patch - placebo tablets
Drug: Placebo patch — Placebo patch designed to match active Climara patches.
  Arms: Placebo patch - Resveratrol tablets; Placebo patch - placebo tablets
Dietary Supplement: Resveratrol
  Arms: Placebo patch - Resveratrol tablets
Dietary Supplement: Placebo — Placebo tablets designed to match active resveratrol tablets.
  Arms: Climara patch - placebo tablets; Placebo patch - placebo tablets

SUMMARY:
This pilot study plans to learn more about the aging of blood vessels and arteries in women. As women age and go through menopause, their risk for cardiovascular disease increases. Also with aging and menopause, levels of the reproductive hormone estradiol decline. Hormone replacement therapy to restore estradiol levels does not protect women from cardiovascular disease, so lifestyle changes, such as regular exercise, are recommended to reduce disease risk. However, there are differences between men and women in their response to exercise. In older men, exercise improves the health of their arteries, but in postmenopausal women, exercise does not provide this benefit. The purpose of this pilot study is to determine whether low estradiol levels in postmenopausal women are responsible for the poor vascular response to exercise. In this study the investigators will also test whether treatment with resveratrol, a plant compound found in red wine, improves postmenopausal women's response to exercise. The investigators hypothesize that acute treatment with estrogen or resveratrol will improve vascular responses to an acute bout of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50-70 and at least 1 year beyond menopause;
* resting blood pressure <140/90 mmHg;
* plasma glucose concentrations <110 mg/dL under fasting conditions;
* BMI < 35;
* LDL cholesterol < 160 mg/dL;
* sedentary or recreationally active (<3 days of vigorous aerobic exercise);
* no use of OCs, HT, or other medications that might influence cardiovascular function;
* nonsmokers;
* no use of vitamin supplements, blood thinners or NSAIDS, or willing to stop use one month prior to and for the duration of the study;
* not taking any other medications that would interact with E2 patch or resveratrol to confound interpretation of results.

Exclusion Criteria:

* history of or active E2-dependent neoplasms, acute liver or gallbladder disease, vaginal bleeding, venous thromboembolism, hypertriglyceridemia (≥ 150 mg/dL), and CVD;
* known allergy to transdermal patch, or resveratrol;
* history of stomach ulcer or bleeding;
* other contraindications to HT or resveratrol.
* other conditions for which individuals will be excluded from the study include: diabetes, active infection, history of seizures or disease that affects the nervous system or an abnormal resting ECG.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie L Moreau, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy women ages 50-70 years, at least 1 year beyond menopause and free of overt cardiovascular or chronic diseases.
Pre-assignment Details: 7 participants did not qualify to participate in the study after consent/enrollment.
Groups:
- Visit 1 Placebo - Visit 2 Estrogen - Visit 3 Resveratrol: Visit 1 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Placebo tablet: Placebo tablets designed to match active resveratrol tablets.
  Visit 2 Estrogen: Climara patch was worn two days prior to and during the exercise visit.
  Placebo tablet:Placebo tablets designed to match active resveratrol tablets.
  Visit 3 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Resveratrol tablet: Resveratrol tablets were given on the morning of the exercise visit.
- Visit 1 Resveratrol - Visit 2 Placebo - Visit 3 Estrogen: Visit 1 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Resveratrol tablet: Resveratrol tablets were given on the morning of the exercise visit.
  Visit 2 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Placebo tablet: Placebo tablets designed to match active resveratrol tablets.
  Visit 3 Estrogen: Climara patch was worn two days prior to and during the exercise visit.
  Placebo tablet:Placebo tablets designed to match active resveratrol tablets.
- Visit 1 Estrogen - Visit 2 Resveratrol - Visit 3 Placebo: Visit 1 Estrogen: Climara patch was worn two days prior to and during the exercise visit.
  Placebo tablet:Placebo tablets designed to match active resveratrol tablets.
  Visit 2 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Resveratrol tablet: Resveratrol tablets were given on the morning of the exercise visit.
  Visit 3 Placebo patch: Placebo patch designed to match active Climara patches and was worn two days prior to exercise visit.
  Placebo tablet: Placebo tablets designed to match active resveratrol tablets.
Period: Overall Study
Arm/Group | Visit 1 Placebo - Visit 2 Estrogen - Visit 3 Resveratrol | Visit 1 Resveratrol - Visit 2 Placebo - Visit 3 Estrogen | Visit 1 Estrogen - Visit 2 Resveratrol - Visit 3 Placebo
Started | 6 | 6 | 6
Completed | 6 | 5 | 4
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Back pain preventing exercise | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Brachial Artery Flow-mediated Dilation at Each Time Point
Description: Brachial artery flow-mediated dilation represents the percent change in artery diameter (before and after blood pressure cuff inflation-deflation) within each time point.
Time Frame: Up to 2 hours post-exercise
Population: Images were considered invalid and removed from analysis if the vascular boundaries were not able to be identified.
Measure: Mean (Standard Error); unit: Percent Change
Groups:
- Placebo Patch - Resveratrol Tablets: Postmenopausal women will be given a placebo patch to wear for two days prior to the exercise visit and a resveratrol tablet (dosed at 250mg) to take the morning of the exercise visit.
  Placebo patch: Placebo patch designed to match active Climara patches.
  Resveratrol
- Climara Patch - Placebo Tablets: Postmenopausal women will be given a transdermal estrogen patch to wear (0.05mg/day) for two days prior to the exercise visit and a placebo tablet to take the morning of the exercise visit.
  Climara
  Placebo: Placebo tablets designed to match active resveratrol tablets.
Arm/Group | Placebo Patch - Placebo Tablets | Placebo Patch - Resveratrol Tablets | Climara Patch - Placebo Tablets
Number analyzed (Participants) | 13 | 12 | 12
Percent Change
  Baseline | 4.11 (0.44) | 6.93 (0.79) | 5.86 (0.65)
  30 min after exercise: number analyzed (Participants) | 13 | 11 | 10
  30 min after exercise | 3.20 (0.45) | 5.88 (0.81) | 5.41 (0.67)
  60 min after exercise: number analyzed (Participants) | 13 | 12 | 10
  60 min after exercise | 3.23 (0.44) | 7.01 (0.79) | 6.99 (0.69)
  120 min after exercise: number analyzed (Participants) | 13 | 11 | 12
  120 min after exercise | 4.35 (0.44) | 7.57 (0.81) | 8.03 (0.65)

2. Secondary Outcome: Gene and Protein Expression in Peripheral Blood Mononuclear Cells
Description: No gene and protein data were analyzed.
Time Frame: baseline, 1-2 hours post-exercise
Population: No data were collected for this outcome measure.
Arm/Group | Placebo Patch - Placebo Tablets | Placebo Patch - Resveratrol Tablets | Climara Patch - Placebo Tablets
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Nitrate/Nitrite Levels
Description: Measure of nitric oxide
Time Frame: baseline, 1-2 hrs post-exercise
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Placebo Patch - Placebo Tablets | Placebo Patch - Resveratrol Tablets | Climara Patch - Placebo Tablets
Number analyzed (Participants) | 15 | 15 | 15
micromolar
  Baseline | 121.3 (57.6) | 134.2 (65.6) | 110.9 (53.5)
  60 min after exercise | 108.6 (48.5) | 109.6 (59.2) | 118.2 (61.1)
  120 min after exercise | 114.7 (54.2) | 118.7 (56.0) | 111.1 (60.6)

ADVERSE EVENTS:
Arm/Group | Placebo Patch - Placebo Tablets | Placebo Patch - Resveratrol Tablets | Climara Patch - Placebo Tablets
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No